## MCC-21-18632

# SUCCEED: Engaging Black Men in CRC Screening

NCT05980182

06/30/2023

# Approved by the VCU IRB on 6/30/2023

### RESEARCH PARTICIPANT INFORMATION SHEET

STUDY TITLE: SUCEED Pilot Project: Engaging Black Men in CRC Screening

VCU INVESTIGATOR: Maria Thomson, PhD,

**VSU INVESTIGATOR:** Larry Keen, PhD

You are invited to participate in a research study about men's health and prevention of colorectal cancer. Your participation is voluntary.

In this study, you will be asked to do the following things:

- 1. Download the SUCCEED App from Pattern Health and complete the consent form
- 2. Complete a brief survey about yourself.
- 3. View the materials on the app.
- 4. Respond to up to 4 texts from the study team
- 5. Complete a follow up survey at 2 and 12 weeks

If you have any questions, concerns, or complaints about this study now or in the future, please contact Dr. Maria Thomson, 804-628-2640, <a href="mailto:maria.thomson@vcuhealth.org">maria.thomson@vcuhealth.org</a>

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Web site at any time.

### WILL I BE PAID TO PARTICIPATE IN THE STUDY?

You will be paid \$30 for each survey completed for a total of up to \$90 if all 3 surveys are completed. Payments will be made by gift card.

### **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. This certificate will offer the protections described here. A Certificate of Confidentiality helps the researchers keep your information private. For example, researchers can refuse to give out your information in a court case. Researchers may have to give your information if the study is audited, or if the information is required by the Food and Drug Administration (FDA).

The researchers cannot prevent you or others, for example a member of your family, from sharing information about you or your involvement in this research. If you give an insurer, employer, or other person permission to receive research information, then the researchers may not use the Certificate to withhold that information.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others.